CLINICAL TRIAL: NCT03163082
Title: Targeting Couple Coercion to Impact Health Behaviors and Regimen Adherence
Brief Title: Couple Interaction and Health Behaviors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Collaborators: National Institute of Dental and Craniofacial Research (NIDCR) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 15-01090; 1UH2DE025980-01 (NIH)
Record Dates: First submitted 2017-05-19; First posted 2017-05-22 (Actual); Last update posted 2020-11-13 (Actual); Status verified 2020-11

CONDITIONS: Couples; Relationship, Marital
Keywords: Coercion theory; Corrosive Couple Coercion
MeSH Terms: interventions — Behavior Therapy

STUDY DESIGN:
Intervention Model Description: Within-subject design over 2 visits.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Cognitive Intervention (Active Comparator): The cognitive intervention has partners come up with reasons why their partners do things they don't like, until they come up with benign attributions for those behaviors.
  Interventions: Other: Cognitive Intervention
- Behavioral Intervention (Active Comparator): The behavioral intervention has partners develop an if-then plan for dealing with conflict and negativity, using strategies to downregulate their own negative emotions.
  Interventions: Behavioral: Behavioral Intervention
- Interpretation Bias (Active Comparator): The Interpretation Bias intervention has partners look at "morphed" facial expressions and determine whether the face is happy or angry. Positive feedback is given for rating the faces as happy and negative feedback is given for rating the faces as angry.
  Interventions: Other: Interpretation Bias
- Evaluative Conditioning (Active Comparator): The Evaluative Conditioning intervention presents partners with pictures of ambiguous adult faces (conditioned stimuli) and pairs them with positive word descriptors (unconditioned stimuli; e.g., generous; loving).
  Interventions: Other: Evaluative Conditioning

INTERVENTIONS:
Other: Cognitive Intervention — The cognitive intervention has partners come up with reasons why their partners do things they don't like, until they come up with benign attributions for those behaviors.
  Arms: Cognitive Intervention
Behavioral: Behavioral Intervention — The behavioral intervention has partners develop an if-then plan for dealing with conflict and negativity, using strategies to downregulate their own negative emotions.
  Arms: Behavioral Intervention
Other: Interpretation Bias — The Interpretation Bias intervention has partners look at "morphed" facial expressions and determine whether the face is happy or angry. Positive feedback is given for rating the faces as happy and negative feedback is given for rating the faces as angry.
  Arms: Interpretation Bias
Other: Evaluative Conditioning — The Evaluative Conditioning intervention presents partners with pictures of ambiguous adult faces (conditioned stimuli) and pairs them with positive word descriptors (unconditioned stimuli; e.g., generous; loving).
  Arms: Evaluative Conditioning

SUMMARY:
The investigators are interested in typical couple interactions and health behaviors. In particular, the investigators are interested in different ways that each partner in a coupled relationship reacts to and understand each other's behavior, and in their health behaviors.

DETAILED DESCRIPTION:
If couples decide to participate in this study, they will come visit the laboratory at a time that is convenient for them.

Couples will be asked to participate in the following activities. These activities will be video recorded and recordings will be kept digitally on a secure password-protected server. Video recordings will be assigned a number, and names and identifying information will not be associated in any way with the video recordings. If couples do not want to be video recorded, they can not participate in this research.

* Upon arrival at the laboratory during both visits, the subject runners will explain the tasks to participants. The subject runners also will measure participants' heart rates and skin moisture. To do so the subject runners will place 9 sensors on each person's body: on the collar bones, the lower left rib cage, the upper and mid-chest, the upper and mid-back, and the palm of their nondominant hand. The sensors will be connected to small machines that participants will carry. Participants will still be able to move freely around the room.
* Partners will be asked to sit separately while they complete a questionnaire that asks about their relationship.
* There will either be:

  * A short discussion where the subject runners will discuss their responses to their partner's behavior or the intentions behind their partner's behavior. A quarter of the research subjects in this study will complete a task where their responses to their partner's behaviors are discussed and another quarter of the subjects will complete a task where the reasons for their partner's behavior are discussed. Which type of discussion they have will be "randomly assigned", which means that a computer will generate this decision before they arrive for their visit.
  * Or a short computerized activity where partners will look at a series of images and descriptions or will be asked to rate a series of images with facial expressions. A quarter of the research subjects in this study will complete a computerized activity where they will look at a series of images and descriptions and another quarter of the subjects will complete a computerized activity where they will rate a series of images with facial expressions. Which type of activity participants have will be "randomly assigned", which means that a computer will generate this decision before they arrive for their visit.
* Couples will complete a video-recorded problem-solving task, where they discuss some of the things that they would like each other to do, do different, or change.
* There will either be:

  * A 10-minute break. Drinks and snacks will be provided during the break.
  * Or a task where partners will rate what they felt and thought during their conversation with their partner while watching a video of their conversation.
* At the end of these activities, the subject runners will provide couples with the opportunity to discuss the visit and any other questions or concerns they may have. They will not be asked to participate in any additional visits or questionnaires after their second visit.

ELIGIBILITY:
Inclusion Criteria:

* Both partners must be 18 years of age or older
* At least one of the partners in the couple dyad carries a Type 2 Diabetes (T2D) diagnosis or is at risk for T2D.
* The couple must qualify on relationship characteristics
* The couple must be married or have lived together for at least 6 months

Exclusion Criteria:

-If individuals do not meet the above criteria, they will be excluded from the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 142 (Actual)
Dates: Start 2017-05-01 (Actual); Primary Completion 2020-06-30 (Actual); Study Completion 2020-06-30 (Actual)

PRIMARY OUTCOMES:
Problem-Solving Task | 20 minutes per visit
  Couples will complete a video-recorded problem-solving task, where they discuss some of the things that they would like each other to do, do different, or change.
Health Behaviors | 10 minutes per visit
  Health Behaviors
Video-Mediated Emotion Recall | 20 Minutes per visit
  The video-mediated recall procedure (Gottman & Levenson, 1985; Lorber, 2007) is a procedure by which parents and/or a member of a couple view a videotape of their interaction with their partner or child. While watching the video, they use a dial to rate their experienced emotion and/or cognitions moment-by-moment during the interaction task. Partners assigned to the interpretation bias and evaluative conditioning interventions will be given this task.

SECONDARY OUTCOMES:
Psychophysiological Measures | 1.5-3 hours per visit
  The investigators also will measure participants' heart rates and skin moisture. To do so the subject runners will place 9 sensors on each person's body: on the collar bones, the lower left rib cage, the upper and mid-chest, the upper and mid-back, and the palm of their nondominant hand. The sensors will be connected to small machines that participants will carry. Participants will still be able to move freely around the room.

CONTACTS AND LOCATIONS:
Overall Officials: Richard Heyman, Principal Investigator — NYU Langone Health
Locations (1):
- New York University School of Medicine, New York, New York, United States

REFERENCES:
- [Derived] Smith Slep AM, Heyman RE, Mitnick DA, Lorber MF, Rhoades KA, Daly KA, Nichols SR, Eddy JM. Do Brief Lab-Based Interventions Decrease Coercive Conflict Within Couples and Parent-Child Dyads? Behav Ther. 2023 Jul;54(4):666-681. doi: 10.1016/j.beth.2023.01.006. Epub 2023 Feb 2. PMID 37330256

DOCUMENTS (1):
  • Informed Consent Form (2018-03-28): https://cdn.clinicaltrials.gov/large-docs/82/NCT03163082/ICF_003.pdf